CLINICAL TRIAL: NCT01336036
Title: Etiology, Clinical Manifestations and Risk Factors for Community-acquired Pneumonia in Patients Admitted to Hospital
Brief Title: Causes and Outcomes of Community Acquired Pneumonia
Acronym: CAP
Status: Completed | Type: Observational
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Responsible Party: Sponsor
Other Study IDs: 03HN
Record Dates: First submitted 2011-04-06; First posted 2011-04-15 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum Blood Urine Nasal and Throat swab
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a descriptive clinical research aiming:

* To describe the clinical spectrum and clinical characteristics of community acquired pneumonia (CAP) in patients admitted to hospital
* To identify the etiology of CAP and the antibiotic sensitivity of the isolated organisms
* To identify the risk factors that influence the severity of CAP

DETAILED DESCRIPTION:
In Vietnam, the range and relative contribution of organisms causing CAP remain unclear, largely because diagnostic tools are limited and clinical research uncommon. An improved understanding of the risk factors, etiology and clinical outcomes of CAP in Vietnam would contribute to improved approaches to patient diagnosis and clinical management. This will be achieved by following the clinical and laboratory progress and treatment outcomes of in-patients diagnosed with CAP from admission to discharge. Comparative analyses will be between subgroups including survivor and non-survivor, severe CAP and non-severe CAP, known etiology and unknown etiology, SIRS, sepsis, severe sepsis and shock septic.

ELIGIBILITY:
Inclusion Criteria:

* Patients > or = 18 years of age
* Patient meets the criteria of pneumonia (below), established within 36h of hospitalization
* Patient is not hospitalized or residing in a long-term-care facility within 14 days before the onset of symptoms
* Patient has not been at a referral hospital for >2 days before admission to the study hospital
* Informed consent to participate in the study is provided

Exclusion Criteria:

* Severe immunosuppression as judged by the enrolling physician (e.g. HIV, leukemia, lymphoma, chemotherapy for solid tumors, long-term corticosteroid use or other immunosuppressive drugs)
* Known active tuberculosis or current treatment for tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 patients with community acquired pneumonia who meet the below inclusion/ exclusion criteria will be recruited at two hospitals in Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are stable at Day 3, 7 and 14 | up to 14 days
  • Criteria for clinical stability
  * Temperature < or = 37.8oC
  * Heart rate < or = 100 beats/min
  * Respiratory rate < or = 24 breaths/min
  * Systolic blood pressure > or = 90 mm Hg
  * Arterial oxygen saturation > or = 90% or pO2 > or = 60 mm Hg on room air
  * Ability to maintain oral intake
  * Normal mental status

SECONDARY OUTCOMES:
Day 14 mortality | 14 days
  Proportion of patients who die at Day 14
Length of stay (days) | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Length of stay from admission to discharge in days
Need for mechanical ventilation | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Length of ventilation time | participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kinh V Nguyen, PhD, Principal Investigator — National Hospital of Tropical Diseases; Peter Horby, Dr., Principal Investigator — Oxford University Clinical Research Unit - Hanoi; Rogier van Doorn, MD, Principal Investigator — Oxford University Clinical Research Unit
Locations (2):
- Vietnam (2):
  - National Hospital of Tropical Diseases, Hanoi, Hanoi
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City

REFERENCES:
- See also: OUCRU studies public site — http://www.oucru.org/index.php?option=com_content&view=article&id=336&mode=0&fil=&ox=&cd=03HN&type=&inv=&en=&vn=&ran=0.41076726020631754